CLINICAL TRIAL: NCT01749137
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of RM-493, a Melanocortin 4 Receptor (MC4R) Agonist in Obese Patients
Brief Title: Phase 2 Study to Evaluate Safety and Efficacy of RM-493 in Obese Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM-493-003
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Overweight
Keywords: Overweight
MeSH Terms: conditions — Overweight | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Setmelanotide (Experimental): Participants received 1 milligram (mg) setmelanotide every day by continuous subcutaneous infusion using the Omnipod insulin pump for a duration of 90 days.
  Interventions: Drug: Setmelanotide
- Placebo (Placebo Comparator): Participants received placebo matching setmelanotide every day by continuous subcutaneous infusion using the Omnipod insulin pump for a duration of 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Setmelanotide — Daily subcutaneous infusion
  Other Names: RM-493
  Arms: Setmelanotide
Drug: Placebo — Daily subcutaneous infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of RM-493 on mean percent body weight loss, and other weight loss parameters as well as Pharmacokinetic (PK) profile, and ambulatory blood pressure in obese participants. The study is designed to evaluate the efficacy and tolerability of a single dose of RM-493. The study drug (RM-493 and placebo) will be administered subcutaneously in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the age of 18 and 65.
2. Able to provide voluntary, written informed consent with comprehension of all aspects of the protocol, prior to any study procedures.
3. In good general health, without significant medical history, physical examination findings, or clinical laboratory abnormalities.
4. Body Mass Index: 35-50 Kg/m^2, inclusive. It is planned that approximately 20 (but no more than 50% of the total participants enrolled) of these participants will have a BMI ≥ 40 Kg/m^2
5. Stable body weight (+/- 5 Kg) during previous 6 months.
6. Blood pressure (<150/95 mmHg); may include stable dose (≥ 30 days of use) of up to two anti-hypertensive medications to achieve control that are intended to remain on a stable dose during the protocol.
7. Willingness and demonstrates ability to self-administer study medication subcutaneously via an infusion pump during the placebo practice period.
8. Willing to maintain a healthy diet and exercise regime throughout study as recommended by counseling at study start.
9. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception from the Screening Period through the completion of study treatment: hormonal, condom with spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intrauterine device (IUD). Hormonal contraception must have started at least 3 months prior to screening. A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception. Participants must agree to practice the above birth control methods for 30 days after completion of study treatment as a safety precaution.
10. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months (and confirmed with a screening follicle stimulating hormone (FSH) level in the post-menopausal range), do not require contraception during the study.
11. Males with female partners of childbearing potential must agree to use two medically acceptable forms of contraception as described above, with one of the two forms being condom with spermicide, from the Screening Period through 90 days after completion of study treatment. Males with female partners of childbearing potential who themselves are surgically sterile (status post vasectomy) must agree to use condoms with spermicide over the same period of time.

Exclusion Criteria:

1. Fasting blood glucose > than 140 mg/dL.
2. Haemoglobin A1c (HbA1c) ≥6.5%.
3. Thyroid stimulating hormone (TSH) level outside the normal range.
4. Creatinine > 1.5 times the upper limit of normal.
5. Liver function tests > 2 times the upper limit of normal.
6. Active or history of any significant medical condition including renal, hepatic, pulmonary, gastrointestinal, cardiovascular, genitourinary, endocrine, immunologic, metabolic, neurologic or hematological disease.
7. Participants with a history of the following:

   1. Uncontrolled hypertension;
   2. Diabetes requiring medical treatment, presently or in the past;
   3. Major depressive disorder within the last 2 years;
   4. Any lifetime history of a suicide attempt;
   5. Any suicidal behavior in the last month;
   6. Other severe psychiatric disorders (e.g. schizophrenia, bipolar disorder, severe eating disorders including bulimia).
8. A patient health questionnaire - 9 (PHQ-9) score of ≥15.
9. Any suicidal ideation of type 4 or 5 on the columbia suicide severity rating scale (C-SSRS).
10. Prior bariatric surgery.
11. Treated with anorectic agents or drugs with anorexia as a frequent side event.
12. Taking 3 or more anti-hypertensive medications.
13. Acute illness or history of illness, which in the opinion of the Investigator, could pose a threat or harm to the participant or obscure interpretation of laboratory test results or interpretation of study data.
14. History of human immunodeficiency virus (HIV) infection.
15. History of significant drug hypersensitivity or anaphylaxis.
16. History of hypersensitivity to proteins (e.g., allergy shots).
17. Any clinically significant abnormalities on screening laboratories as determined by the Investigator.
18. Abnormal 12-lead electrocardiogram (ECG) at screening or pre-dose (Day 1), except minor deviations deemed to be of no clinical significance by the Investigator. QTc must be < 450 ms.
19. Received any experimental drugs or devices or have participated in a clinical study within 30 days prior to dosing.
20. Hospitalization for surgery within the 3 months prior to screening except for minor outpatient procedures, or any planned hospitalizations during the study period.
21. Poor venous access or inability to tolerate venipuncture.
22. Inability to attend all study visits or comply with protocol requirements including fasting and restrictions on concomitant medication intake.
23. Participation in weight loss programs during the study period, including nutritional supplements/ replacements other than as recommended by nutritional counseling provided at study start.
24. Use of prescription medications on a regular basis with the following exceptions:

    1. Contraceptives (must be on for ≥3 months);
    2. Hormone replacement therapy (must be on stable dose for ≥3 months);
    3. Antihypertensives (<3 medications on a stable dose for ≥ 30 days);
    4. Statins (dose must be ≤ half the maximum dose; must be on a stable dose ≥3 months);
    5. Fibrates (must be on stable dose for ≥3 months);
    6. Niacin (must be on stable dose for ≥3 months);
    7. Thyroxin (stable dose for ≥ 30 days);
    8. The last use of any other prescription medication must have been greater than 5 half-lives for the specific medication or at least 14 days prior to randomization, whichever is longer.
25. Women who are pregnant or are breast feeding.
26. Previously randomized and dosed in this study or previously exposed to RM-493.
27. History of alcohol or drug abuse within 5 years of Screening Visit.
28. Any other reason, which in the opinion of the Investigator would confound proper evaluation of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2013-09-28 (Actual); Study Completion 2013-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Miami, Florida
  - Lexington, Kentucky
  - Rochester, New York
  - Raleigh, North Carolina
  - Dallas, Texas
  - Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Setmelanotide | Placebo
Started | 37 | 37
Completed | 22 | 26
Not Completed | 15 | 11
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 8 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all randomized participants with both a baseline and at least one post-dose efficacy observation (for at least one efficacy endpoint).
Groups:
- Setmelanotide: Participants received 1 mg setmelanotide every day by continuous subcutaneous infusion using the Omnipod insulin pump for a duration of 90 days.
- Total: Total of all reporting groups
Arm/Group | Setmelanotide | Placebo | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (9.77) | 40.4 (11.72) | 41.2 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 35 | 66
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 16 | 31
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 113.65 (16.074) | 111.20 (10.031) | 112.43 (13.362)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight
Description: The mean percent change from baseline in body weight at Day 90 was analyzed.
Time Frame: Baseline and Day 90
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 33 | 36
Percent change | -2.0 (2.82) | -0.3 (2.96)
Statistical Analysis 1: Comparison: Setmelanotide vs Placebo; Test type: Superiority — P-value from a mixed-effects analysis of covariance model with treatment, visit and visit-by-treatment interaction as factors, baseline weight as a covariate, and participant as the random effect; p = 0.059, Mixed Model Repeated Measures (MMRM); Treatment Difference = -1.1, 95% CI 2-sided [-2.27 to 0.04], Standard Error of Mean 0.58

2. Secondary Outcome: Change From Baseline in Body Weight
Description: The mean change from baseline in body weight at day 90 was analyzed.
Time Frame: Baseline and Day 90
Population: FAS population with available data specified time point.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 33 | 36
Kilograms | -2.2 (3.39) | -0.3 (3.34)
Statistical Analysis 1: Comparison: Setmelanotide vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.079, MMRM; Treatment Difference = -1.2, 95% CI 2-sided [-2.48 to 0.14], Standard Error of Mean 0.66

3. Secondary Outcome: Percentage of Participants Who Lost ≥ 5% of Their Baseline Body Weight
Description: The percentage of participants who lost ≥ 5% of their baseline body weight was analyzed. 95% confidence interval is calculated based on Clopper-Pearson.
Time Frame: Baseline up to Day 90
Population: FAS population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 33 | 36
percentage of participants | 9.1 [1.9 to 24.3] | 5.6 [0.7 to 18.7]
Statistical Analysis 1: Comparison: Setmelanotide vs Placebo; Test type: Superiority; p = 0.513, Cochran-Mantel-Haenszel — P-values from a Cochran-Mantel-Haenszel (CMH) test, controlling for site and the stratification factor severely obese (yes/no)

4. Secondary Outcome: Number of Participants Who Consistently Achieved Targeted Plasma Concentration of ~6 Nanogram Per Milliliter (ng/mL)
Description: Number of Participants Who Consistently Achieved Targeted Plasma Concentration of ~6 ng/mL were reported.
Time Frame: Day 1: pre-dose and 2-hours post-infusion, Day 7, 14, 28, 56, and 90
Population: The pharmacokinetic population included all participants who received any of the study drug infusion and have at least one post-dose safety assessment and who had evaluable plasma concentrations for RM-493.
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 37
Participants | 8

5. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An adverse event (also referred to as an adverse experience) could be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. A treatment-emergent AE was defined as an AE with an onset date on or after day 1.
Time Frame: From first dose of study drug (Day 1) until end of study (Up to 184 days)
Population: The Safety Analysis Set consisted of all participants who received any of the study drug infusion and had at least one post-dose safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 37 | 37
percentage of participants | 75.7 | 48.7

6. Secondary Outcome: Change From Baseline in Ambulatory Blood Pressure Monitoring Parameter (ABPM) - Systolic Blood Pressure
Description: Summary of individual average data at daytime, nighttime and 24 hours was reported.
Time Frame: Baseline and Day 28
Population: ABPM Completers population as participants who had both baseline and post-baseline assessment of ABPM parameters
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 13 | 12
millimeter of mercury (mmHg)
  Daytime individual average | -2.45 (14.071) | 1.83 (12.200)
  Night time individual average | -3.26 (13.310) | 1.24 (10.721)
  24 hour (hr) individual average | -2.79 (13.174) | 1.61 (11.165)

7. Secondary Outcome: Change From Baseline in ABPM - Diastolic Blood Pressure
Description: Summary of individual average data at daytime, nighttime and 24 hours was reported.
Time Frame: Baseline and Day 28
Population: ABPM Completers
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 13 | 12
mmHg
  Daytime individual average | -1.62 (9.672) | 1.39 (5.591)
  Night time individual average | -0.96 (9.586) | 0.60 (5.184)
  24 hr individual average | -1.38 (9.261) | 1.09 (4.977)

8. Secondary Outcome: Change From Baseline in ABPM - Mean Arterial Blood Pressure
Description: Summary of individual average data at daytime, nighttime and 24 hours was reported.
Time Frame: Baseline and Day 28
Population: ABPM Completers.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 13 | 12
mmHg
  Daytime individual average | -1.27 (10.886) | 1.70 (8.056)
  Night time individual average | -2.15 (10.589) | 0.86 (6.536)
  24 hr individual average | -1.65 (10.205) | 1.38 (7.018)

9. Secondary Outcome: Change From Baseline in ABPM - Heart Rate
Description: Summary of individual average data at daytime, nighttime and 24 hours was reported.
Time Frame: Baseline and Day 28
Population: ABPM Completers.
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 13 | 12
Beats per minute (BPM)
  Daytime individual average | 1.44 (6.861) | -1.90 (8.702)
  Night time individual average | -0.28 (8.293) | 0.05 (10.420)
  24 hr individual average | 0.70 (6.703) | -1.07 (8.242)

10. Secondary Outcome: Change From Baseline in ABPM - Pulse Pressure
Description: Summary of individual average data at daytime, nighttime and 24 hours was reported.
Time Frame: Baseline and Day 28
Population: ABPM Completers.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 13 | 12
mmHg
  Daytime individual average | -0.83 (6.320) | 0.44 (8.060)
  Night time individual average | -2.30 (6.038) | 0.65 (6.820)
  24 hr individual average | -1.41 (5.655) | 0.52 (7.366)

11. Secondary Outcome: Percent Change From Baseline in Body Weight in Severely Obese Participants
Description: The mean percent change from baseline in body weight in severely obese participants at Day 90 was analyzed.
Time Frame: Baseline and Day 90
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 17 | 17
Percent change | -2.3 (3.34) | -0.7 (3.08)
Statistical Analysis 1: Comparison: Setmelanotide vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.387, MMRM; Treatment Difference = -0.8, 95% CI 2-sided [-2.50 to 0.98], Standard Error of Mean 0.87

12. Secondary Outcome: Percentage of Participants Who Lost ≥ 5% of Their Baseline Body Weight in Severely Obese Participants
Description: The percentage of participants who lost ≥ 5% of their baseline body weight loss in severely obese participants was analyzed. 95% confidence interval is calculated based on Clopper-Pearson confidence interval.
Time Frame: Baseline up to Day 90
Population: FAS population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide | Placebo
Number analyzed (Participants) | 17 | 17
percentage of participants | 11.8 [1.5 to 36.4] | 11.8 [1.5 to 36.4]
Statistical Analysis 1: Comparison: Setmelanotide vs Placebo; Test type: Superiority; p = 1.000, Cochran-Mantel-Haenszel — P-values from a Cochran-Mantel-Haenszel (CMH) test, controlling for site

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) until end of study (Up to 184 days)
Description: Safety Population
Arm/Group | Setmelanotide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/37
Other Adverse Events (participants affected / at risk) | 28/37 | 18/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Setmelanotide (N=37) | Placebo (N=37)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Setmelanotide (N=37) | Placebo (N=37)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (5)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Infusion site infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 2 (2) | 0 (0)
Application site dermatitis (General disorders) | 1 (1) | 0 (0)
Application site erosion (General disorders) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 1 (1) | 0 (0)
Application site haemorrhage (General disorders) | 0 (0) | 1 (1)
Application site pain (General disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 5 (5) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Infusion site discolouration (General disorders) | 1 (2) | 0 (0)
Infusion site pruritus (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Dark circles under eyes (Eye disorders) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Gum discoloration (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.